CLINICAL TRIAL: NCT05130645
Title: Evaluation of Mandibular Mental Angle and Mandibular Profile Angle in Prediction of Difficult Intubation and Comparison With Other Tests
Brief Title: Evaluation of Mandibular Mental Angle and Mandibular Profile Angle
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Sule Ozdemir, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: Mentum angle
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mental Angle — In order to standardize and measure the mental angle, the projection of the mental will be accepted as the midline, the jaw structure will be transferred to the paper using the profile contour meter, and the angle between the angulus mandible and the mental will be measured and recorded with a digital protractor.
  Other Names: Profiler Type Mental Angle

SUMMARY:
Airway management is extremely important for providing safe anesthesia. Endotracheal intubation, on the other hand, is the most important step in airway management, especially since it requires rapid and successful execution. Inadequate airway management; is associated with complications that require high-level care and cost, such as death, brain damage, increased need for intensive care, prolonged recovery period, and emergency tracheostomy. 15-25% of anesthesia-related deaths are associated with airway management. 17% of settled cases against anesthesiologists are composed of airway-related events (often difficult intubation, inadequate oxygenation/ventilation, and pulmonary aspiration).

An important point in ensuring airway patency is preoperative evaluation. Difficulties arising from anatomical features can be revealed by careful evaluation of mouth opening, the structure of tongue and palate, thyromental distance (TMM), sternomental distance (SMM), mobility of cervical vertebrae, jaw occlusion, and necessary precautions can be taken.

The most commonly used tests to determine the degree of difficulty of intubation are the modified Mallampati test, the thyromental distance, the upper lip bite test, the inter incisor space, and the sternomental distance. Recent studies are trying to confirm the sensitivity and specificity of existing tests. However, there is no test with 100% specificity and sensitivity in predicting difficult laryngoscopy and intubation.

DETAILED DESCRIPTION:
In this prospective observational study, two new parameters "mandibular profile angle" and "mandibular mental angle" will be evaluated with the Cormack-Lehane Score during laryngoscopy as a predictor of difficult laryngoscopy. Modified Mallampati test, neck circumference, thyromental distance, sternomental distance, and many other tests have been used for predicting difficult intubation however, none of them are able to predict "difficult intubation" exactly. "mandibular profile angle" and "mandibular mental angle" may provide new horizons for predicting difficult intubation. These two measurements will be compared with the Cormack-Lehane score during laryngoscopy for sensitivity, specificity, and positive or negative predictive values. As well as the Cormack-Lehane Score, we will be comparing these angle measurements' predictive values with the other specified predictive tests such as Modified Mallampati test, neck circumference, thyromental distance, sternomental distance.

Having received informed consent, 1000 ASA I-III patients aged between 18-80, who will be operated under general anesthesia, will be included in this prospective observational study. The number of patients is determined according to the numbers in previous studies, but will be finalized as 90% power and 5% error as a result of the power analysis after the prior study.

Before the anesthesia induction the Modified Mallampati test, neck circumference, thyromental distance, sternomental distance will be measured as well as "mandibular profile angle" and "mandibular mental angle". "Mandibular profile angle" is defined as; The angle between the mentum of the mandibula and the lateral tips of the mandibula where the profiler ends. "Mandibular mental angle" is defined as; the angle between the mentum of the mandibula and the two ends of the mandibular arch.

After induction of anesthesia, the difficulty of laryngoscopy will be determined by Cormack-Lehane Score by a senior anesthesiologist.

Having received the measurements, tests for sensitivity and specificity, and negative/positive predictive values for difficult intubation will be processed.

ELIGIBILITY:
Inclusion Criteria:

* General Anesthesia
* ASA I,II,III

Exclusion Criteria:

* Patients with upper respiratory tract tumors
* history of surgery, burns and trauma to the upper respiratory tract
* congenital head-neck anomaly,
* giant goiter, and
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will operated under general anesthesia by endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-28 (Estimated); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Mandibular mental angle to predict the degree of difficulty in intubation | 5 min before intubation
  The angle between the mentum of the mandibula and the lateral tips of the mandibula where the profiler ends
Mandibular profile angle to predict the degree of difficulty in intubation | 5 min before intubation
  "Mandibular mental angle" is defined as; the angle between the mentum of the mandibula and the two ends of the mandibular arch.

SECONDARY OUTCOMES:
Cormack- Lehane grading system | Procedure (During the use of direct laryngoscopy for intubation)
  It will be measured by an anesthesiologist during the use of direct laryngoscopy during intubation
Modified Mallampati test | 5 min before intubation
  The modified Mallampati test (MMT) is based on the visibility of the pharyngeal structures by opening the mouth as much as possible and sticking out the tongue while the patient is in a sitting position and the head is in a neutral position.
Neck circumference | 5 min before intubation
  Neck circumference is measured using a tape measure at the level of the thyroid cartilage with the head in a neutral position.
Thyromental distance | 5 min before intubation
  The thyromental distance is found by measuring the distance between the mental prominence of the mandible and the thyroid cartilage when the patient's head is in full extension.
Sternomental distance | 5 min before intubation
  Sternomental distance, when the patient's head is in full extension; It is determined by measuring the distance between the upper border of the manbrium sterni and the mental prominens of the mandible.
Upper lip bite test | 5 min before intubation
  The upper lip bite test is found by measuring the degree of biting the upper lip with the lower incisors.
Evaluation of mouth opening | 5 min before intubation
  It is found by measuring the distance between the upper and lower anterior incisors when the mouth is at its maximum opening.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Şule Özdemir, Study Chair — Diskapi Yildirim Beyazit ERH

IPD SHARING:
Plan to Share IPD: Undecided
If we can take a permission to share